CLINICAL TRIAL: NCT00101439
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Period, Crossover Study to Evaluate the Effects of Ezetimibe on the Postprandial Lipoprotein Response in Patients With Primary Hypercholesterolemia
Brief Title: A Study to Evaluate the Effects of Ezetimibe (MK-0653) on the Postprandial (Following a Meal) Lipoprotein Response in Participants With Primary Hypercholesterolemia (High Cholesterol) (MK-0653-072)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-072; MK-0653-072; 2005_001
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: Primary Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe→Placebo (Experimental): After a 2-week single- blind placebo run-in, participants will receive ezetimibe 10 mg once daily for 4 weeks and then receive placebo once daily for 4 weeks.
  Interventions: Drug: ezetimibe; Drug: Comparator: placebo
- Placebo→ Ezetimibe (Experimental): After a 2-week single- blind placebo run-in, participants will receive placebo once daily for 4 weeks and then receive ezetimibe10 mg once daily for 4 weeks.
  Interventions: Drug: ezetimibe; Drug: Comparator: placebo

INTERVENTIONS:
Drug: ezetimibe
  Other Names: MK-0653
Drug: Comparator: placebo

SUMMARY:
A study to evaluate the cholesterol-lowering effects of ezetimibe in participants with primary hypercholesterolemia (high cholesterol) after eating a meal that is high in cholesterol. The primary hypothesis is that treatment with ezetimibe 10 mg/day reduces the cholesterol concentration of the chylomicron-containing Sf≥400 fraction following a cholesterol-enriched test meal.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be otherwise healthy men and women (if not on oral contraceptives or hormone replacement therapy) 18 through 70 years of age with moderately high cholesterol.

Exclusion Criteria:

* Individuals on other lipid-lowering therapy (medicines that lower cholesterol) including statins (within 6 weeks) and fibrates (within 8 weeks) prior to administration of the study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-11-10 (Actual); Primary Completion 2006-10-24 (Actual); Study Completion 2006-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Ezetimibe→Placebo | Placebo→ Ezetimibe
Started | 28 | 30
Completed | 28 | 30
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Ezetimibe→Placebo | Placebo→ Ezetimibe
Started | 28 | 30
Completed | 28 | 28
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe→Placebo | Placebo→ Ezetimibe | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (8.84) | 48.4 (9.48) | 49.7 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 22 | 28 | 50

OUTCOME MEASURES:

1. Primary Outcome: Total Cholesterol Concentration of Chylomicron (Sf≥400) Fractions After a Cholesterol-Rich Test Meal
Description: On each of 2 days prior to the last day of each treatment period, participants consumed 2 large eggs in the evening. On the morning of the final day of each treatment period, fasting participants were given a site-prepared, cholesterol-enriched milkshake that provided 1114 calories of total energy (~44% of calories from fat, ~40% of calories from carbohydrate and ~17% of calories from protein) and 504 mg of cholesterol. The milkshake was consumed over a 15-minute period. Plasma samples were collected immediately prior to consumption of the test meal (baseline) and at 2, 3, 4, and 6 hours afterwards for isolation and analysis of lipoprotein fractions. The geometric mean concentration level was calculated using data obtained at all timepoints.
Time Frame: Immediately prior to consumption of the test meal (baseline) and at 2, 3, 4, and 6 hours after test meal on Day 28 of each treatment period.
Population: Participants who received at least one dose of study drug and did not have any protocol violations.
Measure: Geometric Mean (Full Range); unit: mg/dL
Groups:
- Ezetimibe: Participants who received ezetimibe 10 mg in active treatment period regardless of randomly assigned sequence
- Placebo: Participants who received placebo in active treatment period regardless of randomly assigned sequence
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 56 | 56
mg/dL | 0.45 [0.10 to 2.82] | 0.50 [0.02 to 1.90]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.241, ANOVA — Data were back-transformed from the log scale and adjusted for treatment; Geometric Mean Ratio (GMR) = 0.89, 95% CI 2-sided [0.73 to 1.08] — GMR=Ezetimibe divided by placebo

2. Secondary Outcome: Total Cholesterol Concentration of Chylomicron-remnant (Sf 60-400) Subfractions After a Cholesterol-Rich Test Meal
Description: On each of 2 days prior to the last day of each treatment period, participants consumed 2 large eggs in the evening. On the morning of the final day of each treatment period, fasting participants were given a site-prepared, cholesterol-enriched milkshake that provided 1114 calories of total energy (~44% of calories from fat, ~40% of calories from carbohydrate and ~17% of calories from protein) and 504 mg of cholesterol. The milkshake was consumed over a 15-minute period. Plasma samples were collected immediately prior to consumption of the test meal (baseline) and at 2, 3, 4, and 6 hours afterwards for isolation and analysis of lipoprotein subfractions. The geometric mean concentration level was calculated using data obtained at all timepoints.
Time Frame: as for outcome 1
Population: Participants who received at least one dose of study drug and did not have any protocol violations.
Measure: Geometric Mean (Full Range); unit: mg/dL
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 56 | 56
mg/dL | 4.87 [1.25 to 23.74] | 4.78 [0.93 to 31.36]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.812, ANOVA — Data were back-transformed from the log scale and adjusted for treatment; Geometric Mean Ratio (GMR) = 1.02, 95% CI 2-sided [0.87 to 1.20] — GMR=Ezetimibe divided by placebo

ADVERSE EVENTS:
Time Frame: up to 10 weeks
Description: All participants who received at least 1 dose of study drug. Adverse events are reported by study drug received at the time of the event and not by treatment sequence.
Groups:
- Ezetimibe: Participants received 10 mg ezetimibe once daily for 4 weeks
- Placebo: Participants received placebo once daily for 4 weeks
Arm/Group | Ezetimibe | Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 0/56 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.